CLINICAL TRIAL: NCT06684509
Title: Using of Atorvastatin for Anthracyclin _ Associated Cardiotoxicity in Hemetological Malignancies Patients.
Brief Title: Atorvaststin and Cardiotoxicity in Acute Myloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mahmoud Abd Rabou, Physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Atorvaststin and cardiotoxicit
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Leukemia; Hodgkin Disease
Keywords: Cardiotoxicity; Atrovastatin
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Cardiotoxicity

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non Atrovastatin group (No Intervention): control group of the same condition they will not tkae atrovastatin
- Atrovastatin group (Experimental): patients will receive atorvaststin 40mg/daily , started before anthracyclin treatment and continued 12 months
  Interventions: Drug: Atrovastain

INTERVENTIONS:
Drug: Atrovastain — atorvaststin 40mg/daily , started before anthracyclin treatment and continued 12 months
  Arms: Atrovastatin group

SUMMARY:
The research proposal focuses on evaluating the efficacy of atorvastatin in reducing cardiotoxicity caused by anthracycline chemotherapy in patients with hematologic malignancies, specifically acute myeloid leukemia (AML) and non-Hodgkin lymphoma (NHL). The study will be conducted at Assiut University Hospitals and will include patients aged 18 or older receiving anthracycline-based treatments (3+7 regimen for AML and CHOP regimen for NHL).

The background highlights that anthracyclines, a class of chemotherapeutic agents, can cause serious side effects, particularly cardiotoxicity. The research aims to investigate whether atorvastatin, a statin used to lower cholesterol, can mitigate this risk by improving cardiac function in patients undergoing chemotherapy.

The study will be a randomized controlled trial with a sample size of 46 participants. It will assess left ventricular ejection fraction (LVEF) as the primary outcome to determine the effect of atorvastatin on reducing cardiotoxicity. Secondary outcomes include identifying high-risk patients and further understanding the impact of atorvastatin.

The study also adheres to ethical guidelines, ensuring patient consent and confidentiality. Data analysis will be performed using IBM SPSS, and results will be disseminated in scientific journals, with support from Assiut Medical School's Grants Office if funding is approved.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years Patient with hematologic malignany ( Acute myeloid leukemia on 3,7 regimen or non-Hodkin Lymphoma on CHOP regimen) Cardiac function with EF ≥60%

Exclusion criteria:

Cardiac dysfunction with EF < 60% Other hematologic malignancies Pregnant women and breastfeeding Patients refuse participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity | During the study period along 12 months
  Effect of atorvaststin for anthracyclin induced cardiotoxicity measured through Echo and ECG

SECONDARY OUTCOMES:
Cardiotoxicity events correlation to high risk patients | along 12 months
  we will correlate cardiotoxicity with the factors that make those patients high risk group for cardiotoxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes